CLINICAL TRIAL: NCT01238354
Title: Conservative Treatment of Obesity at Røros Rehabilitation Centre - A Randomised Trial
Brief Title: Family & Friends - the Significance of a Significant Other in Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RSSO-2010/2
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Obesity
Keywords: Weight Loss; Social support
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without friend (Active Comparator): Being in the weight loss programme without friend or family member
  Interventions: Behavioral: Without friend
- With friend (Experimental): Having the friend or family member stay together with the patient for 2-3 days for every 3 week stay at the clinic in the weight loss programme
  Interventions: Behavioral: With friend

INTERVENTIONS:
Behavioral: With friend
  Arms: With friend
Behavioral: Without friend
  Arms: Without friend

SUMMARY:
This study focuses on the difficulties to maintain a weight loss and behavioural change after having been in a institutional intermittent weight loss programme.

We explore if including a member of the family or a close friend in the treatment influences weight loss maintenance after completion of the programme.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity
* 18-50 years of age
* Having a relative or close friend who is willing to participate

Exclusion Criteria:

* Pregnancy
* Serious mental illness
* Severe overeating behaviour
* Significant reduced physical functioning
* Having undergone bariatric surgery earlier
* Serious heart disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maintenance of weight loss | 2 years after termination of programme

CONTACTS AND LOCATIONS:
Overall Officials: Bård Kulseng, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Roros Rehabiliteringssenter, Røros, Norway

IPD SHARING:
Plan to Share IPD: Undecided